CLINICAL TRIAL: NCT07163052
Title: Hemodynamic Evaluation of Left Atrial Pressure in Relationship to Pulmonary Capillary Wedge Pressure in Cardio Thoracic Patients
Acronym: HEART
Status: Not yet recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Ufuk Baldan, Resident cardiac surgery, MD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: HEART
Record Dates: First submitted 2025-08-24; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Cardiogenic Shock; Pulmonary Edema Cardiac Cause
Keywords: LV unloading; post-cardiotomy shock; PCS; filling pressures
MeSH Terms: conditions — Shock, Cardiogenic; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Total cohort: Patients with and without LV unloading under different cardiac indeces via cardiopulmonary bypass

SUMMARY:
Accurate hemodynamic monitoring is critical in cardiothoracic surgery, where left atrial pressure (LAP) serves as the gold standard for assessing left-sided cardiac filling pressures. However, its invasive nature limits use, favoring pulmonary capillary wedge pressure (PCWP) via Swan-Ganz catheter as a surrogate. Despite widespread use, evidence on their agreement under dynamic conditions-such as varying cardiac index (CI) flows during cardiopulmonary bypass (CPB) or left ventricular (LV) unloading-remains inconsistent and unstudied in adult cardiac surgery.

Existing data show conflicting correlations: one study found that PCWP 35% higher than LAP in non-surgical patients, and another study found closer alignment in specific cohorts. This knowledge gap carries clinical urgency, as decisions on pulmonary edema management, vasopressor use, and LV decompression rely on these measurements.

Building on Laplace's law, we hypothesize that LV unloading reduces ventricular wall stress (afterload), lowering myocardial oxygen demand and altering the LAP-PCWP relationship. Elevated CI during CPB may further distort this interaction via increased pulmonary-left atrial pressure gradients.

The primary objective is to determine if PCWP reliably reflects LAP under standard CI-flow (2.4 L/min/m²) without unloading, using Bland-Altman analysis (±5 mmHg clinical margin). Secondary objectives assess agreement at other CI levels (1.8-2.6 L/min/m²), LV unloading effects, and patient/surgical variable impacts.

DETAILED DESCRIPTION:
Effective hemodynamic monitoring is essential for optimizing postoperative management in cardiothoracic surgery. Left atrial pressure (LAP) is considered the gold standard for assessing left-sided cardiac filling pressures, but is typically measured directly only in selected cases due to its invasive nature. Pulmonary capillary wedge pressure (PCWP), measured via a Swan-Ganz catheter, is widely used as a less invasive surrogate for LAP. However, evidence suggests that the agreement between PCWP and directly measured LAP may vary under different hemodynamic conditions, particularly at higher cardiac index (CI) flow rates and with or without left ventricular (LV) unloading. To date, no in-vivo study has systematically quantified the agreement between these two methods in adult patients during cardiopulmonary bypass (CPB) at varying flow rates and unloading conditions.

Existing studies report inconsistent correlations between LAP and PCWP. For example, one study observed PCWP values 35% higher than LAP in non-surgical patients, while another study noted tighter correlations in specific cohorts. However, no in-vivo data exist for adult cardiac surgery patients under controlled CI-flow rates (+/- LV unloading). This gap is clinically critical, as decisions regarding pulmonary edema management, vasopressor use, and LV decompression rely on these measurements.

Building on Laplace's law, we hypothesize that LV unloading reduces ventricular wall stress (afterload), thereby lowering myocardial oxygen demand and improving recovery. Computational models and animal studies suggest that unloading decreases LV end-diastolic pressure (LVEDP) and left atrial (LA) volume, which may alter the LAP-PCWP relationship. Elevated CI during CPB could further modulate this interaction, as increased flow rates may exacerbate pressure gradients between the pulmonary vasculature and left atrium.

The primary objective of our study is therefore to determine whether PCWP can be considered an adequate surrogate for directly measured LAP under standard CI-flow (2.4 L/min/m²) without LV unloading, using a Bland-Altman analysis. Secondary objectives include evaluating the agreement between LAP and PCWP at other CI-flow rates and with LV unloading, as well as exploring the influence of patient characteristics and surgical variables. By addressing these questions, we hope to provide evidence to guide the interpretation of PCWP in clinical practice, potentially improving the safety and outcomes of patients undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* the primary procedure is cardiac surgery by median sternotomy
* the use of CPB
* patients undergoing aortic valve replacement (AVR) due to aortic regurgitation, mitral valve plasty (MVP), mitral valve repair (MVR), valve sparing aortic root replacement or supracoronary aorta ascendens replacement (SCAR)
* left ventricular ejection fraction of 60% or more
* no clinical or echocardiographic signs of preoperative decompensation cordis
* only elective procedures

Exclusion Criteria:

* patients with left ventricular hypertrophy (LVH), severe aortic stenosis or hypertrophic obstructive cardiomyopathy. LVH is defined as an increased LVMI greater than 95 grams per square meter (g/m²) in women and greater than 115 g/m² in men.
* patients with echocardiographically observed RV or LV dilatation are assessed using specific criteria. For RV dilatation, a TAPSE of less than 14 millimeters or an RV FAC of less than 35% is indicative of dilatation. For LV dilatation, an LV end-diastolic (LVED) diameter greater than 2.7 centimeters per square meter or exceeding 117% of the predicted value, adjusted for age and body surface area, is considered dilated.
* patients undergoing more than one type of procedure (i.e. double valve surgery, CABG and AVR)
* postoperative aortic valve mean pressure gradient of more than 20 mm Hg and mitral valve mean pressure gradient of more than 5 mm Hg
* postoperative paravalvular leak grade 2 or more
* postoperative persistent regional wall abnormalities or electrocardiographic signs of acute ischemia
* other significant valve pathology, such as moderate mitral regurgitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective cardiac surgery for aortic valve regurgitation, mitral valve, coronary or aortic disease. We aim to include patients without significant impairment in cardiac function. Nonetheless, there are inherent primary and secondary effects of cardiac pathology leading to structural disease. The procedures, as noted in the inclusion criteria (4.2), are standard procedures in our hospital and are regularly performed. We want to select the patient from our wait list. No extra measures are taken to include the patients.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Agreement between left atrial pressure (LAP) and pulmonary capillary wedge pressure (PCWP) under standard cardiac index (CI) conditions. | Intraoperatively
  The primary outcome is the mean absolute difference between LAP and PCWP, quantified using Bland-Altman analysis. PCWP will be considered an adequate surrogate for LAP if the 95% limits of agreement fall within ±5 mmHg.
  Independent: cardiac index fixed at 2.4 L/min/m² without LV unloading Dependent: difference between LAP and PCWP (mmHg)

SECONDARY OUTCOMES:
Effect of different cardiac index (CI) flow rates and LV unloading on agreement between left atrial pressure (LAP) and pulmonary capillary wedge pressure (PCWP) | Intraoperatively
  Agreement between LAP and PCWP will be assessed for each CI flow rate and LV unloading condition using Bland-Altman analysis (95% limits of agreement). Correlation between LAP and PCWP will also be calculated (Pearson or Spearman) (mmHg)
Pre- and postoperative changes in left atrial pressure (LAP) and pulmonary capillary wedge pressure (PCWP) in mitral valve patients | Intraoperatively
  Comparison of LAP and PCWP before and after mitral valve surgery. Statistical analysis will be performed using paired t-test or Wilcoxon Signed-Rank test, depending on data distribution (mmHg).
Association between echocardiographic parameters and invasive pressure measurements: LVEDV | Intraoperatively
  Echocardiographic chamber volumes (LVEDV) will be summarized (mean ± SD or median [IQR]) and associated with LAP/PCWP. Used for pressure-volume loop construction with invasive pressures.
  mL
Association between echocardiographic parameters and invasive pressure measurements: LV wall thickness | Intraoperatively
  LV hypertrophy will be recorded and associated with LAP/PCWP.
  mm
Association between echocardiographic parameters and invasive pressure measurements: LVEF | Intraoperatively
  Functional measures of LV and RV performance, diastolic filling pressures, and mitral regurgitation severity will be summarized and associated with LAP/PCWP.
  LVEF: %
Association between echocardiographic parameters and invasive pressure measurements: E/e' | Intraoperatively
  Functional measures of leftsided diastolic filling pressures will be summarized and associated with LAP/PCWP.
  E/e' ratio: unitless
Association between echocardiographic parameters and invasive pressure measurements: TAPSE | Intraoperatively
  Functional measures of RV performance will be summarized and associated with LAP/PCWP.
  TAPSE: mm
Association between echocardiographic parameters and invasive pressure measurements: mitral regurgitation grade | Intraoperatively
  Functional measures of mitral regurgitation severity will be summarized and associated with LAP/PCWP.
  Mitral regurgitation: ordinal grade (1-4)
Association between echocardiographic parameters and invasive pressure measurements: LAVI | Intraoperatively
  Echocardiographic chamber volumes (LAVI) will be summarized (mean ± SD or median [IQR]) and associated with LAP/PCWP. Used for pressure-volume loop construction with invasive pressures.
  mL/m²
Association between echocardiographic parameters and invasive pressure measurements: RAVI | Intraoperatively
  Echocardiographic chamber volumes (RAVI) will be summarized (mean ± SD or median [IQR]) and associated with LAP/PCWP. Used for pressure-volume loop construction with invasive pressures.
  mL/m²
Association between echocardiographic parameters and invasive pressure measurements: LVOT dimensions | Intraoperatively
  LVOT dimensions will be recorded and associated with LAP/PCWP.
  mm

IPD SHARING:
Plan to Share IPD: No